CLINICAL TRIAL: NCT04696263
Title: Prospective Single-Center Randomized Study Of Single-Port Versus Multi-Port Robotic Radical Prostatectomy
Brief Title: Single-Port Versus Multi-Port Robotic Radical Prostatectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closure based on study population not found and not enough study staff
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE7820
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Malignant Neoplasm of Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Extraperitoneal SinglePort (SP) Robotic Radical Prostatectomy (Da Vinci ® SP system) (Active Comparator): All participants will undergo SOC robotic radical prostatectomy.
  The procedure for this arm uses the Da Vinci ® SP system. Access point consists of one 3.5 cm single infraumbilical incision for the SP-RARP
  Interventions: Device: Da Vinci ® SP system - SP Robotic Radical Prostatectomy
- Extraperitoneal MultiPort (MP) Robotic Radical Prostatectomy (Da Vinci ® Xi system) (Active Comparator): All participants will undergo SOC robotic radical prostatectomy.
  The procedure for this arm uses the Da Vinci ® Xi system, where four 8mm trocars will be used along with a 12 mm assistant trocar (a surgical instrument) to create six small incisions during the surgery
  Interventions: Device: Da Vinci ® Xi system - MP Robotic Radical Prostatectomy

INTERVENTIONS:
Device: Da Vinci ® Xi system - MP Robotic Radical Prostatectomy — After pneumoperitoneum is established, four 8mm, one 12 mm, and one 5 mm trocars are placed for instrumentation. After the robot is docked, radical prostatectomy is performed with the SOC approach.
  Arms: Extraperitoneal MultiPort (MP) Robotic Radical Prostatectomy (Da Vinci ® Xi system)
Device: Da Vinci ® SP system - SP Robotic Radical Prostatectomy — After induction of general anesthesia and supine participant positioning, a 3.5 cm infraumbilical incision will be made for single-port access into the space of Retzius. Radical prostatectomy is then performed with the SOC approach
  Arms: Extraperitoneal SinglePort (SP) Robotic Radical Prostatectomy (Da Vinci ® SP system)

SUMMARY:
The purpose of this study is to compare two different techniques to perform the standard of care surgery to treat prostate cancer. This surgery is called robotic radical prostatectomy. There are two robotic surgical systems approved by the Food and Drug Administration (FDA) to perform this surgery. First system is called the Da Vinci ® Xi system. With this system, six small incisions are made during the surgery. Second system is called the Da Vinci ® SP system. With this system a single incision is made during the surgery. Same surgery is done with each surgical system. This study aims to understand whether a single incision surgery ends up with better recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed prostate cancer, stage T1a, T2a or T2b prostate cancer using MRI staging.
* Life expectancy greater than 10 years.
* Participants must have ability to understand and the willingness to sign a written informed consent document or have a surrogate with the ability to understand and the willingness to sign a written informed consent for radical prostatectomy.

Exclusion Criteria:

* Participants with any prior extensive pelvic surgery or pelvic fractures.
* Prior treatment for prostate cancer such as radiotherapy or focal therapy.
* Uncorrected coagulopathy.
* Active soft tissue or urinary infection.
* Poor surgical risk (defined as American Society of Anesthesiology score > 3)
* Any condition or history of illness or surgery that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient (e.g. significant cardiovascular conditions that significantly affect the life expectancy, chronic opiate use, pain syndrome, or drug abuse.)
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Recovery of Urinary Continence Following Catheter Removal | Up to 12 months post-treatment
  Continence will be defined as the absence of pads (even safety pads).

SECONDARY OUTCOMES:
Operative time | During operation, an average operative time is 192 minutes
  Time elapsed from skin incision to placement of the final skin suture
Estimated blood loss in milliliters | During operation, an average operative time is 192 minutes
  Estimated blood loss, measured in volume (mL)
Number of additional ports | Within 24 hours of surgery
  Number of additional ports needed in surgery
Number of SP procedures converted to other procedure types | Within 24 hours of surgery
  For SP procedures, conversion to MP robotic surgery or standard laparoscopic surgery, or open surgery will be recorded
Intraoperative complication rate | Within 24 hours of surgery
  Intraoperative complication rate compared between the two systems
Number of participants requiring Intraoperative Trendelenburg position | Within 24 hours of surgery
  Intraoperative Trendelenburg position requirement for the participant will be recorded. Position involves placing the head low and feet elevated, increasing blood return to the heart, cardiac output and vital organ perfusion
Intraoperative peritoneum breach rate | Within 24 hours of surgery
  Intraoperative peritoneum breach rate as defined by intraoperative pneumoperitoneum after insufflation of extraperitoneal space
Visual analog pain scale scores | Within 7 days of surgery
  Pain intensity will be evaluated with a visual analog pain scale, a validated instrument scored from 0 to 10, 10 being the worst
Units of parenteral morphine equivalents (mg) | Up to 1 month post-procedure
  Analgesic requirements will be obtained from medical charts and reported as units of parenteral morphine equivalents (mg)
Time to liquid oral intake | Post-surgery, an average of 16 hours
  Time to liquid oral intake
Time to solid oral intake | Post-surgery, an average of 16 hours
  Time to solid oral intake
Number of postoperative complications | Within 30 days
  Postoperative complications recorded according to the Clavien- Dindo classification
Body image questionnaire scores | Up to 1 year
  Body image perception, measured using the body image questionnaire, which consists of two sub-scales: the body image scale, which assesses attitudes to bodily appearance and consists of five questions (score 5-20) where higher scores mean worse outcomes, and the cosmetic scale which assesses the degree of satisfaction with the appearance of the scar and consists of three questions (score 3-24), where higher scores mean worse outcomes.
Participant and Observer Scar Assessment Scale scores | Up to 1 year
  Scar evaluation by using a validated assessment tool, the Participant and Observer Scar Assessment Scale.17 It consists of two scales: the observer scale and the participant scale (Figs. 1 and 2). Both scales contain six items that are scored numerically. Each of the six items on both scales has a 10-step score, with 10 indicating the worst imaginable scar or sensation. The total score of both scales consists of adding the scores of each of the six items (range, 6 to 60). The lowest score, 6, reflects normal skin, whereas the highest score, 60, reflects the worst imaginable scar.
Number of pads used daily | Up to 1 year
  Urinary continence, assessing the number of pads used daily. Continence will be defined as the absence of pads (even safety pads)
International Index of Erectile Function (IIEF-5) scale scores | Up to 1 year
  Erectile Function assessed by the IIEF-5 scale, consisting of 5 questions, with scores ranging from 5-25. 25 being great and 5 being the worst
Time to return-to-work | Up to 1 year
  Time to return-to-work, reported in days
Time to baseline | Up to 1 year
  Time to baseline defined as the amount of time between surgery and when the patient becomes pain free and does not need painkillers
Hospital stay in hours | Post-surgery, an average of 16 hours
  Hospital stay, counted in hours from the time of transfer to the post anesthesia care unit (PACU) to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Kaouk, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This trial will not study a drug, device, biological/vaccine, radiation, genetic, combination product or diagnostic test